CLINICAL TRIAL: NCT02432521
Title: Predictors of Treatment Response of Motor Sequels After a Cerebrovascular Accident
Brief Title: Predictors of Treatment Response of Motor Sequels After a Stroke
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Linamara Rizzo Battistella, MD PhD, Full Professor, Medical School of the University of Sao Paulo, Post Graduate Program in Medical Sciences of the Medical School of the University of Sao Paulo, University of Sao Paulo General Hospital
Other Study IDs: 35583814.1.0000.0068_CAAE
Record Dates: First submitted 2015-04-16; First posted 2015-05-04 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Cerebrovascular Accident
Keywords: stroke; transcranial magnetic stimulation (TMS); Electroencephalography (EEG); Cerebrovascular Accident; Brain Vascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Conventional rehabilitation program from IMREA — The IMREA rehabilitation program lasts about 18 weeks and consists of two weekly sessions of 60 minutes of physical therapy, occupational therapy, as well as weekly sessions of speech therapy, nursing, nutrition, psychology and social work. Conventional therapies are typically composed of stretching and strengthening exercises both upper and lower limbs, mobilizations, functional training. The only fact that differ the subjects from the protocol from the patients from the IMREA Institute are the clinical and neurophysiological evaluations that will be performed before and after the end of the conventional rehabilitation program previously described.

SUMMARY:
The cerebrovascular accident (CVA) is currently the leading cause of death in Brazil and it is estimated that there are about 62 million stroke survivors worldwide. Thus, the stroke sequels are a major public health problem not only in Brazil but in the world, with existing treatments often insufficient for complete recovery. Thus this study aims to identify predictors of different responses from rehabilitation therapy through the evaluation of clinical and neurophysiological data performed before and after treatment. For the neurophysiological study will be used the association of electroencephalogram (EEG) and transcranial magnetic stimulation (TMS). This last one will be performed in the baseline and after a single Transcranial direct current stimulation (tDCS) session, aiming to leverage the ability of those technics to analyze the cerebral plasticity. As a secondary objective: 1) Identify specific features of brain plasticity involved in recovery from stroke and discuss the possible implications of these findings in the therapeutic approach; 2) Search possible electrophysiological markers that can be used as surrogate outcome of stroke of motor sequel.

DETAILED DESCRIPTION:
The cerebrovascular accident (CVA) is currently the leading cause of death in Brazil and it is estimated that there are about 62 million stroke survivors worldwide. Thus, the stroke sequels are a major public health problem not only in Brazil but in the world, with existing treatments often insufficient for complete recovery. Thus, the search for new treatments is necessary, as well as the need to optimize and individualize the existing treatments. Several approaches are being used in order to find predictors of the recovery of patients after the stroke, highlighting the most recent studies using magnetic resonance imaging (MRI) with tractography. However these studies have important limitations such as high cost, but mainly the low capacity of this technique to quantify brain plasticity known to play an important role in the recovery of stroke sequelae. Thus, techniques to measure brain plasticity theory offer the best potential to predict the resilience of post stroke injury, among which stands out transcranial magnetic stimulation (TMS).

TMS is a noninvasive brain stimulation techniques suitable for measuring the motor cortex excitability which in turn is used as an indirect measure of brain plasticity. Another interesting approach is the combination of TMS with the study of neuronal function through the electroencephalogram (EEG). The EEG under the stroke, has also been suggested as sequelae recovery predictor, however in this scenario the association of these findings with TMS has not yet been explored. Thus this study aims to identify predictors of different responses from rehabilitation therapy through the evaluation of clinical and neurophysiological data performed before and after treatment. For the neurophysiological study will be used the association of electroencephalogram (EEG) and transcranial magnetic stimulation (TMS). This last one will be performed in the baseline and after a single Transcranial direct current stimulation (tDCS) session, aiming to leverage the ability of those technics to analyze the cerebral plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis (Functional magnetic Resonance (FMR) and/or Computerized tomography (TC) ) of the stroke;
* More than one month from the date of the stroke;
* Clinical stability;
* Signed and dated informed consent form.

Exclusion Criteria:

* Disturbs that forbid the adherence in treatment;
* Subjects already undergoing in other researches;
* Pregnant women;
* Lesions that could affect the proposed therapy;
* The occurence of lesion or muscle,joint pain that could forbid the therapy;
* Destabilization of the clinical comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of hemiplegia ambulatory from the Institute of Physical Medicine and Rehabilitation (IMREA) from the Clinics Hospital (HC) of the Medical School of the University of Sao Paulo (USP)
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in motor cortex excitability as measured by Transcranial magnetic stimulation (TMS) | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
  A noninvasive brain stimulation techniques suitable for measuring the motor cortex excitability
Change in spontaneous electrical brain activity as assessed by Electroencephalogram (EEG) | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
  The record of the brain's spontaneous electrical activity

SECONDARY OUTCOMES:
cinematic variables analyzed with robotic | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
  speed, acceleration, articular angulation, time-to-point, task execution time, target displacement
Mini-mental State Examination | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Visual Analog Scale of Pain | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Verbal fluency test | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Boston naming test | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Hamilton Rating scale of depression | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
The Kinesthetic and visual imagery questionnaire (KVIQ) | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
National Institutes of Health Stroke Scale (NIHSS) | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Stroke Impact Scale (SIS) | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Von Frey test | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Functional Independence Measure | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Epworth Sleepiness Scale | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Fugl-Meyer Assessment | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Medical Research Council Scale | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Modified Ashworth Scale | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Finger Tapping | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Jebsen-Taylor Hand Function Test | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline
Purdue Pegboard test | At baseline, 11th week, 22nd week, and after 3 and 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Linamara Battistella, Md PhD, Principal Investigator — Head Professor, Medical School of the University of Sao Paulo, pos graduation program at the Medical Science of the Medical School of the University of Sao Paulo
Locations (1):
- Centro de Pesquisa Clínica do Instituto de Medicina e Reabilitação do HCFMUSP, São Paulo, Brazil

REFERENCES:
- [Background] Norrving B, Kissela B. The global burden of stroke and need for a continuum of care. Neurology. 2013 Jan 15;80(3 Suppl 2):S5-12. doi: 10.1212/WNL.0b013e3182762397. PMID 23319486
- [Background] Stinear C. Prediction of recovery of motor function after stroke. Lancet Neurol. 2010 Dec;9(12):1228-1232. doi: 10.1016/S1474-4422(10)70247-7. Epub 2010 Oct 27. PMID 21035399